CLINICAL TRIAL: NCT06460948
Title: Characterizing Oxytocin Response to Oral Estrogen Administration in Adults With Arginine Vasopressin Deficiency
Brief Title: Identifying Oxytocin Deficiency in Adults With Pituitary Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Elizabeth Austen Lawson (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Austen Lawson, Associate Professor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P001090
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Arginine Vasopressin Deficiency; Oxytocin Deficiency
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic | interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study Model description: In this open-labeled, interventional pilot trial, 16 adults with arginine-vasopressin deficiency and 16 healthy controls balanced for age, sex, and body mass index will be recruited
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arginine-vasopressin deficiency (Experimental): Norethindrone Acetate-Ethinyl Estradiol will be given to participants with arginine-vasopressin deficiency
  Interventions: Drug: Norethindrone Acetate-Ethinyl Estradiol
- Healthy control (Experimental): Norethindrone Acetate-Ethinyl Estradiol will be given to the healthy controls.
  Interventions: Drug: Norethindrone Acetate-Ethinyl Estradiol

INTERVENTIONS:
Drug: Norethindrone Acetate-Ethinyl Estradiol — Estrogen-progestin will be given to participants in both cohorts, arginine-vasopressin deficiency cohort and healthy control cohort.
  Other Names: Estrogen-progestin

SUMMARY:
This is an open-label, pilot study, to characterize oxytocin response to a single dose of oral Estrogen-progestin in patients with arginine-vasopressin deficiency compared to healthy controls. The association between oxytocin levels and measures of psychopathology (i.e., anxiety and depression) and quality of life across groups will be examined. We hypothesize that:

1. Salivary and blood oxytocin response to Estrogen-progestin will be lower in arginine-vasopressin deficiency compared to healthy control.
2. Lower salivary and blood oxytocin levels will be associated with more severe symptoms of anxiety, depression, and social emotional difficulties as well as lower quality of life.

ELIGIBILITY:
Inclusion Criteria:

* AVD Group:

Adults 18-65 years old Arginine-vasopressin deficiency Stable pituitary hormone replacement

* Healthy Control Group Adults 16-65 years old

Exclusion Criteria for all participants:

* History of pulmonary embolism, deep vein thrombosis, breast/endometrial cancer, stroke, transient ischemic attack, myocardial infarction, angina pectoris, or peripheral artery disease
* Pregnancy or breastfeeding within last 8 weeks
* Any significant illness or condition that the investigator determines could interfere with study participation, data collection, or safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in peripheral oxytocin concentration from 0 to 24 hours | Time points: time 0 min (baseline) and 24 hours
  Change in peripheral oxytocin concentration from 0 to 24 hours

SECONDARY OUTCOMES:
Area under the curve of salivary oxytocin from baseline to 48 hours following Estrogen-progestin administration in patients with arginine-vasopressin deficiency compared to healthy controls | From time 0 min (baseline) to 48 hours
  Difference from baseline to oxytocin peak (blood and saliva) between patients with arginine-vasopressin deficiency compared to healthy controls.
  Correlation between oxytocin area under the curve and psychopathology and quality of life measures across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No